CLINICAL TRIAL: NCT02516111
Title: Comparative Evaluation of Autologous PRF, 1% Alendronate and 1.2% Atorvastatin Gel in Treatment of 2/3-walled Intrabony Defects in Chronic Periodontitis Subjects: a Randomized Controlled Clinical Trial
Brief Title: Comparison of Autologous PRF, 1% Alendronate and 1.2% Atorvastatin Gel in Chronic Periodontitis Treatment
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Government Dental College and Research Institute, Bangalore (Other)
Responsible Party: Principal Investigator, Dr. A R Pradeep, Professor and Head, Government Dental College and Research Institute, Bangalore
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GDCRI/ACM/PG/PhD/2/2013-2014M
Record Dates: First submitted 2015-08-03; First posted 2015-08-05 (Estimated); Last update posted 2015-08-05 (Estimated); Status verified 2015-08

CONDITIONS: Chronic Periodontitis
MeSH Terms: conditions — Chronic Periodontitis | interventions — Prolactin-Releasing Hormone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Open flap debridement group (Active Comparator): SRP with Open flap debridement (OFD) alone for treating intrabony defect
  Interventions: Procedure: Open flap debridement (OFD)
- PRF group (Active Comparator): SRP with Open flap debridement (OFD) with autologous Platelet rich fibrin (PRF) placement into intrabony defect
  Interventions: Biological: OFD with PRF
- Alendronate group (Active Comparator): SRP with Open flap debridement (OFD) with 1% Alendronate (ALN) placement into intrabony defect
  Interventions: Drug: OFD with ALN
- Atorvastatin group (Active Comparator): SRP with Open flap debridement (OFD) with 1.2% Atorvastatin (ATV) placement into intrabony defect
  Interventions: Drug: OFD with ATV

INTERVENTIONS:
Procedure: Open flap debridement (OFD) — Oral prophylaxis followed by Open flap debridement (OFD)
  Arms: Open flap debridement group
Biological: OFD with PRF — Oral prophylaxis followed by Open flap debridement (OFD) with Platelet rich fibrin (PRF) placement into the bone defect
  Arms: PRF group
Drug: OFD with ALN — Oral prophylaxis followed by Open flap debridement (OFD) with 1% ALN gel placement into the bone defect
  Arms: Alendronate group
Drug: OFD with ATV — Oral prophylaxis followed by Open flap debridement (OFD) with 1.2% ATV gel placement into the bone defect
  Arms: Atorvastatin group

SUMMARY:
The present study is designed as a single-centre, randomized, controlled clinical trial to evaluate and compare the clinical efficacy of autologous PRF, 1% alendronate (ALN) and 1.2% atorvastatin (ATV) gel placement with open flap debriedement in treatment of intrabony defects in patients with chronic periodontitis.

DETAILED DESCRIPTION:
Background: Platelet-rich fibrin (PRF) is a second-generation platelet concentrate which releases various growth factors that promote tissue regeneration. Alendronate and Atorvastatin are known to inhibit osteoclastic bone resorption and were proposed to have osteostimulative properties by causing osteoblast differentiation in vivo and in vitro as shown by an increase in matrix formation. The aim of the present study is to evaluate and compare the efficacy of autologous PRF, 1% alendronate and 1.2% atorvastatin gel placement with open flap debriedement in treatment of intrabony defects in patients with chronic periodontitis.

Methods: 120 CP subjects with IBD ≥3 mm deep and probing depth (PD) ≥5 mm, following scaling and root planing (SRP), were categorized into four treatment groups: 1) OFD 2) OFD with PRF 3) OFD with 1% ALN gel and 4) OFD with 1.2% ATV gel. Clinical parameters including site specific plaque index (PI), modified sulcus bleeding index (mSBI), probing depth (PD) and relative attachment level (RAL) as well as percentage radiographic intrabony defect depth reduction (DDR) were recorded at baseline before surgery and 9 months post-operatively.

ELIGIBILITY:
Inclusion Criteria:

* Systemically healthy patients with PDs ≥5mm or CALs ≥4 to 6mm and vertical bone loss ≥3 mm on intraoral periapical radiographs with no history of periodontal therapy or use of antibiotics in the preceding 6 months were included

Exclusion Criteria:

* Patients with a known systemic disease
* Known or suspected allergy to the ALN/ bisphosphonates or ATV/statin group
* On systemic ALN/ bisphosphonates or ATV/statin group
* With aggressive periodontitis
* Who used tobacco in any form
* Alcoholics
* Immunocompromised patients
* And pregnant or lactating females were excluded from the study

Ages: 30 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 120 (Actual)
Dates: Start 2014-09; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
defect depth reduction (DDR) | Change from baseline to 9 months

SECONDARY OUTCOMES:
change in clinical attachment level (CAL) | Change from baseline to 9 months
change in probing pocket depths (PPD) | Change from baseline to 9 months
change in plaque index (PI) | Change from baseline to 9 months